CLINICAL TRIAL: NCT00313157
Title: Rate Control in Atrial Fibrillation
Acronym: RATAF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asker & Baerum Hospital (Other)
Responsible Party: Principal Investigator, Sara Reinvik Ulimoe, MD, Asker & Baerum Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-004221-26
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Metoprolol; Diltiazem; Verapamil; Carvedilol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Metoprolol (Active Comparator): Treatment with Metoprolol 100 mg x 1 for three weeks
  Interventions: Drug: Metoprolol
- Diltiazem (Active Comparator): Treatment with Diltiazem 360 mg x 1 for three weeks
  Interventions: Drug: Diltiazem
- Verapamil (Active Comparator): Treatment with Verapamil 240 mg x 1 for three weeks
  Interventions: Drug: Verapamil
- Carvedilol (Active Comparator): Treatment with Carvedilol 25 mg x 1 for three weeks
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Metoprolol
  Other Names: Selo-Zok
  Arms: Metoprolol
Drug: Diltiazem
  Other Names: Cardizem
  Arms: Diltiazem
Drug: Verapamil
  Other Names: Isoptin Retard
  Arms: Verapamil
Drug: Carvedilol
  Other Names: Kredex
  Arms: Carvedilol

SUMMARY:
The purpose of this study is to compare the effect of metoprolol, verapamil, diltiazem and carvedilol on ventricular rate, working capacity and quality of life in patients with chronic atrial fibrillation.

DETAILED DESCRIPTION:
This is a randomised, single blinded, cross-over study comparing the efficacy of metoprolol 100 mg o.d., verapamil 240 mg o.d., diltiazem 360 mg o.d. and carvedilol 25 mg o.d. in reducing ventricular rate in atrial fibrillation. A total of 60 patients will be included, with a minimum of 20 women.Patients will receive each of the drug regimens in a random sequence. Each regimen will be administered for 3 weeks, ensuring that steady-state drug concentration will be attained and to provide an adequate washout of the previous treatment. Following each regimen, exercise ECG and Holter registration will be performed and patients will undergo laboratory evaluation and complete QoL-forms. They will then be started on the next randomly assigned treatment regimen, until the entire sequence of treatment schedules is completed.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or permanent atrial fibrillation with ventricular rate > 80/min at rest and/or > 100/min average at daytime.
* Male or female, age > 18.

Exclusion Criteria:

* Hypersensitivity or contraindication to metoprolol, verapamil, diltiazem or carvedilol.
* Coronary heart disease or heart failure
* Systolic blood pressure < 100 mmHg
* AV-conduction disturbance
* Severe hepatic or renal dysfunction
* Thyrotoxicosis
* Ongoing treatment with Digitalis
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Ventricular rate | Three weeks
  Ventricular rate evaluated after three weeks on study drug treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sara Reinvik Fagertun, MD, Principal Investigator — Asker and Baerum Hospital
Locations (1):
- Vestre Viken Hospital Trust, Baerum Hospital, Rud, Akershus, Norway

REFERENCES:
- [Derived] Horjen AW, Ulimoen SR, Enger S, Norseth J, Seljeflot I, Arnesen H, Tveit A. Troponin I levels in permanent atrial fibrillation-impact of rate control and exercise testing. BMC Cardiovasc Disord. 2016 May 4;16:79. doi: 10.1186/s12872-016-0255-x. PMID 27142292
- [Derived] Corino VD, Sandberg F, Platonov PG, Mainardi LT, Ulimoen SR, Enger S, Tveit A, Sornmo L. Non-invasive evaluation of the effect of metoprolol on the atrioventricular node during permanent atrial fibrillation. Europace. 2014 Nov;16 Suppl 4:iv129-iv134. doi: 10.1093/europace/euu246. PMID 25362163
- [Derived] Ulimoen SR, Enger S, Norseth J, Pripp AH, Abdelnoor M, Arnesen H, Gjesdal K, Tveit A. Improved rate control reduces cardiac troponin T levels in permanent atrial fibrillation. Clin Cardiol. 2014 Jul;37(7):422-7. doi: 10.1002/clc.22281. Epub 2014 Apr 3. PMID 24700386